CLINICAL TRIAL: NCT01139021
Title: A Phase 3, Open-Label, Multi-Center, Extension Study of V72P13E1 to Assess Antibody Persistence at One Year After a Fourth Dose Boost or Two Catch-Up Doses of Novartis Meningococcal B Recombinant Vaccine Administered Starting at 12 Months of Age and to Evaluate the Response to a Third Dose Boost or Two Catch-Up Doses Starting at 24 Months of Age
Brief Title: One Year Antibody Persistence After a Fourth Dose Boost or Two Catch-Up Doses of Novartis Meningococcal B Recombinant Vaccine Administered Starting From 12 Months of Age and Response to a Third Dose Boost or Two Catch-Up Doses Starting at 24 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P13E2; EudraCT No 2009-018101-52
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Meningococcal Disease
Keywords: Children; Meningococcal disease; Prevention; Vaccination
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- B246_12_M12 (Experimental): Subjects assessed one year post administration of rMenB+OMV NZ and MMRV at 12th month after primary vaccination at 2nd ,4th and 6th months of age.
  Interventions: Biological: rMenB+OMV NZ
- B246_12M13 (Experimental): Subjects assessed one year post administration of rMenB+OMV NZ at 12th month and MMRV at 13th month after primary vaccination at 2nd ,4th and 6th months of age.
  Interventions: Biological: rMenB+OMV NZ
- B13_15_27 (Experimental): Subjects assessed at 12 months after two catch-up doses of rMenB+OMV NZ administered to children at 13th and 15th months of age and MMRV at 12th month; at 1 month and 6 months post booster dose administered at 27 months of age.
  Interventions: Biological: rMenB+OMV NZ
- B12_14_26 (Experimental): Subjects assessed at 12 months after two catch-up doses of rMenB+OMV NZ administered to children at either 12th and 14th months of age and MMRV at 12th month; at 1 month and 6 months post booster dose administered at 26 months of age.
  Interventions: Biological: rMenB+OMV NZ
- B_24_26 (Experimental): Subjects assessed at 1 month and 6 months post two catch-up doses of rMenB+OMV NZ administered to naive children at 24 and 26 months of age.
  Interventions: Biological: rMenB+OMV NZ
- B12M13 (Experimental): Subject was randomized in group B13_15_27 but treated as group B12_M13.
  Interventions: Biological: rMenB+OMV NZ

INTERVENTIONS:
Biological: rMenB+OMV NZ — Subjects will be assigned to a study group based on the group assignment in the parent study (follow-on subjects). In addition, one group of naïve age-matched subjects will be recruited at the same study sites. Subjects who had received 4 doses of rMenB+OMV NZ will have one visit including one blood draw. Subjects who had received two catch-up doses in V72P13E1 will receive a third dose boost and will have 3 blood samples drawn. Naïve subjects will receive two catch-up doses and have 3 blood samples drawn.

SUMMARY:
One year antibody persistence after the fourth dose boost or two catch-up doses administered starting from 12 months of age and to evaluate the response to a a third dose boost or two catch-up dose starting at 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children, 23 to 27 months of age (naïve children)
* Available for all the visits scheduled in the study;
* For whom parent(s)/legal guardian(s) have given written informed consent according to local regulations after the nature of the study has been explained;
* Available for all the visits scheduled in the study;
* In good health as determined by medical history, physical examination, clinical judgment of the investigator.
* Healthy children who participated in the immunogenicity part of V72P13E1 and have received their last vaccination 12 months (-30/+60 days) before enrolment in V72P13E2;
* Who received all vaccinations with rMenB+OMV NZ in V72P13 and V72P13E1 according to the protocols;
* Who provided at least the blood sample one month after their fourth dose of rMenB+OMV NZ (groups B246_12M12/B246_12M13) or after their second dose of rMenB+OMV NZ (groups B13_15_27/B12_14_26) in V72P13E1 according to the protocol;
* For whom parent(s)/legal guardian(s) had given written informed consent after the nature of the study has been explained;
* In good health as determined by medical history, physical examination, clinical judgment of the investigator.

Exclusion Criteria:

* Subjects whose parent(s)/legal guardian(s) were unwilling or unable to give written informed consent to participate in the study;
* History of any meningococcal B vaccine administration;
* Previous ascertained or suspected disease caused by N. meningitidis;
* For whom parent(s)/legal guardian(s) have given written informed consent according to local regulations after the nature of the study has been explained;
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
* Antibiotics treatment within 6 days prior to enrolment;
* Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis;
* Any serious chronic or progressive disease
* Known or suspected impairment/ alteration of the immune system,
* Receipt of, or intent to immunize with another vaccine, within 30 days prior and after vaccination with the investigational vaccines (within 14 days for licensed flu vaccines)
* Significant acute or chronic infection within the previous 7 days or axillary temperature ≥38C within the previous day;
* Family members and household members of research staff;
* Any serious chronic or progressive disease according to the judgment of the investigator (e.g., neoplasm, diabetes mellitus Type I, cardiac disease, hepatic disease, neurological disease or seizure, either associated with fever or as part of an underlying neurological disorder or syndrome, autoimmune disease, Human Immunodeficiency Virus (HIV) infection or Acquired Immune Deficiency Syndrome (AIDS), or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition);
* Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids within 30 days prior to enrolment (use of low or moderate doses of inhaled steroids is not an exclusion);
* Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 90 days prior to enrolment;
* Participation in another clinical trial within 90 days prior to enrolment or planned for during study;
* Receipt of, or intent to immunize with any other vaccine(s) within 30 days prior to enrolment (exception: flu-vaccines should not be administered within 14 days prior to enrolment);
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 23 Months to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 508 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Czechia (3):
  - amostatná ordinace praktického lékaře pro děti a dorost Jindřichův Hradec, Hradec
  - Dětské oddělení nemocnice Náchod, Náchod
  - Dětské oddělení nemocnice Pardubice, Pardubice
- Finland (16):
  - University of Tampere Medical School, Vaccine Research Center Tampere, Biokatu 10, Pirkanmaa
  - Espoo Vaccine Research Clinic,, Espoo
  - Helsinki East, Vaccine Research Clinic,, Helsinki
  - Helsinki South, Vaccine Research Clinic,, Helsinki
  - Järvenpää, Vaccine Research Clinic, Jarvenpaa
  - Kokkola Vaccine Research Clinic, Kokkola
  - Kotka Vaccine Research Clinic, Kotka
  - Kuopio Vaccine Research Clinic, Kuopio
  - Lahti Vaccine Research Clinic, Lahti
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
  - Vantaa East, Vaccine Research Clinic, Vantaa
  - Vantaa West, Vaccine Research Clinic, Vantaa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Finland and Czech Republic study center.
Pre-assignment Details: The eligible subjects from V72P13E1 (NCT00847145) who originally participated in the open-label, immunogenicity subset of parent study V72P13 (NCT00657709) and a naïve group, at 24 months of age, who did not previously participate in V72P13 (or V72P13E1) were enrolled in this study.
Groups:
- B246_12M12: Subjects assessed one year post administration of rMenB+OMV NZ and MMRV at 12th month after primary vaccination at 2nd ,4th and 6th months of age.
Period: Overall Study
Arm/Group | B246_12M12 | B246_12M13 | B13_15_27 | B12_14_26 | B_24_26 | B12M13
Started | 152 | 153 | 67 | 19 | 116 | 1
Completed | 151 | 153 | 67 | 18 | 107 | 1
Not Completed | 1 | 0 | 0 | 1 | 9 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B246_12M12 | B246_12M13 | B13_15_27 | B12_14_26 | B_24_26 | B12M13 | Total
Number analyzed (Participants) | 152 | 153 | 67 | 19 | 116 | 1 | 508
Age, Continuous [Mean (Standard Deviation); unit: months] | 25 (1.0) | 25.3 (0.9) | 27.3 (0.9) | 26.6 (1.2) | 24.7 (1.4) | 26 (0) | 25.4 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 68 | 37 | 9 | 61 | 0 | 262
  Male | 65 | 85 | 30 | 10 | 55 | 1 | 246
Region of Enrollment [Number; unit: Number of Subjects]
  Czech Republic | 105 | 113 | 47 | 14 | 66 | 0 | 345
  Finland | 47 | 40 | 20 | 5 | 50 | 1 | 163

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) to Assess Antibody Persistence at 12 Months After a Booster Dose of rMenB+OMV NZ Vaccination.
Description: To assess the immunogenicity in terms of human Serum Bactericidal Assay (hSBA) GMTs through antibody persistence at 12 months after a booster (fourth) dose of Novartis Meningococcal B Recombinant Vaccine (rMenB+OMV NZ) in groups that received a three-dose primary series at 2, 4,6 months of age. Group B246_12M12 received Measles, Mumps, Rubella, Varicella (MMRV) at 12 months of age (concomitantly) and group B246_12M13 received MMRV at 13 months of age (separately).
  Analysis was done on Modified Intention-To-Treat (MITT) population- (Primary).
Time Frame: 12 months post booster (fourth) vaccination.
Population: Analysis was done on Modified Intention-To-Treat (MITT) population (Primary).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- B246_12Tot: Subjects assessed one year post administration of rMenB+OMV NZ at 12th month and MMRV at 12th or 13th month after primary vaccination at 2nd ,4th and 6th months of age
Arm/Group | B246_12M12 | B246_12M13 | B246_12Tot
Number analyzed (Participants) | 147 | 153 | 300
Titers
  H44/76-SL (N=147,152,299) | 7.38 [5.55 to 9.83] | 8.3 [6.17 to 11] | 6.5 [5.63 to 7.5]
  5/99 (N=147,151,298) | 68 [52 to 91] | 90 [67 to 121] | 81 [71 to 94]
  NZ98/254 | 1.57 [1.24 to 1.99] | 1.79 [1.4 to 2.29] | 1.91 [1.7 to 2.15]
  M10713 (N=143,148,291) | 4.37 [3.24 to 5.9] | 3.62 [2.65 to 4.94] | 3.35 [2.88 to 3.9]

2. Primary Outcome: Percentage of Subjects With hSBA ≥1:5 and hSBA ≥1:8 to Assess Antibody Persistence at on 12 Months After a Booster Dose of rMenB+OMV NZ Vaccination.
Description: To assess the immunogenicity in terms of percentage of subjects with hSBA ≥1:5 and hSBA ≥1:8 through antibody persistence at 12 months after a booster (fourth) dose of rMenB+OMV NZ in groups that received a three-dose primary series at 2, 4, 6 months of age. Group B246_12M12 received MMRV at 12 months of age (concomitantly) and group B246_12M13 received MMRV at 13 months of age (separately).
  Analysis was done on MITT population (Primary).
Time Frame: 12 months post booster (fourth) vaccination.
Population: Analysis was done on MITT population (Primary).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B246_12M12 | B246_12M13 | B246_12Tot
Number analyzed (Participants) | 147 | 153 | 300
Percentage of subjects
  H44/76-SL (hSBA ≥1:5) (N=147, 152, 299) | 60 [51 to 68] | 64 [56 to 71] | 62 [56 to 67]
  5/99 (hSBA ≥1:5) (N=147, 151, 298) | 96 [91 to 98] | 99 [95 to 100] | 97 [95 to 99]
  NZ98/254 (hSBA ≥1:5) | 18 [12 to 25] | 17 [11 to 24] | 17 [13 to 22]
  M10713 (hSBA ≥1:5) (N=143, 148, 291) | 40 [32 to 48] | 32 [25 to 41] | 36 [31 to 42]
  H44/76-SL (hSBA ≥1:8) (N=147, 152, 299) | 44 [35 to 52] | 47 [39 to 55] | 45 [39 to 51]
  5/99 (hSBA ≥1:8) (N=147, 151, 298) | 96 [91 to 98] | 98 [94 to 100] | 97 [94 to 99]
  NZ98/254 (hSBA ≥1:8) (N=147, 153, 300) | 12 [7 to 19] | 14 [9 to 21] | 13 [10 to 18]
  M10713 (hSBA ≥1:8) (N=143, 148, 291) | 31 [23 to 39] | 24 [17 to 31] | 27 [22 to 33]

3. Primary Outcome: Geometric Mean Concentrations (GMCs) to Assess Antibody Persistence at One Year After a Booster Dose of rMenB+OMV NZ Vaccination.
Description: To assess the immunogenicity in terms of GMCs determined by Enzyme Linked Immunosorbent Assay (ELISA) through antibody persistence at one year after a booster (fourth) dose of rMenB+OMV NZ in groups that received a three-dose primary series at 2, 4, 6 months of age. Group B246_12M12 received MMRV at 12 months of age (concomitantly) and group B246_12M13 received MMRV at 13 months of age (separately) against vaccine antigen 287-953.
  Analysis was done on MITT population (Primary).
Time Frame: 12 months post booster (fourth) vaccination.
Population: Analysis was done on MITT population (Primary).
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration IU/mL
Arm/Group | B246_12M12 | B246_12M13 | B246_12Tot
Number analyzed (Participants) | 148 | 153 | 301
Concentration IU/mL | 360 [293 to 442] | 389 [314 to 482] | 352 [317 to 391]

4. Secondary Outcome: GMTs to Assess Antibody Persistence at 12 Months After Two Catch-up Doses and 6 Months After Booster Dose of rMenB+OMV NZ Vaccination.
Description: To assess the immunogenicity in terms of hSBA GMTs at 12 months after two catch up doses previously administered to children at either 12 and 14 or 13 and 15 months of age and 6 months after a booster dose of rMenB+OMV NZ administered at 26 or 27 months of age.
  Both the groups received MMRV at 12 months of age.
Time Frame: 12 months post two catch-up dose vaccination and 6 months post booster dose.
Population: Analysis was done on MITT population (Secondary).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- B12+B13Tot: Subjects assessed at 12 months after two catch-up doses of rMenB+OMV NZ administered to children at either 13th and 15th months or 12th and 14th months of age and MMRV at 12th month; at 1 month and 6 months post booster dose administered at 27th or 26th months of age.
Arm/Group | B13_15_27 | B12_14_26 | B12+B13Tot
Number analyzed (Participants) | 67 | 18 | 85
Titers
  H44/76-SL (12months) | 14 [9.01 to 23] | 8.4 [4.13 to 17] | 10 [8 to 13]
  5/99 (12months) (N= 67, 18, 85) | 73 [43 to 123] | 71 [32 to 154] | 65 [49 to 85]
  NZ98/254 (12months) (N= 67, 18, 85) | 1.67 [1.09 to 2.55] | 1.2 [0.64 to 2.27] | 1.75 [1.39 to 2.2]
  M10713 (12months) (N= 64, 18, 82) | 3.74 [2.14 to 6.54] | 3.29 [1.43 to 7.56] | 3.4 [2.5 to 4.61]
  H44/76-SL (6months) (N= 67, 17, 84) | 68 [41 to 113] | 70 [32 to 151] | 51 [38 to 68]
  5/99 (6months) (N= 67, 17, 84) | 524 [332 to 827] | 525 [263 to 1047] | 518 [405 to 664]
  NZ98/254 (6months) (N= 67, 17, 84) | 8.87 [5.23 to 15] | 16 [7.13 to 35] | 8.8 [6.63 to 12]
  M10713 (6months) (N= 66, 16, 82) | 30 [18 to 49] | 36 [17 to 78] | 26 [20 to 33]

5. Secondary Outcome: Percentage of Subjects With hSBA ≥1:5 and hSBA ≥1:8 to Assess Antibody Persistence at 12 Months After Two Catch up Doses and 6 Months After a Booster Doses of rMenB+OMV NZ Vaccination.
Description: To assess the immunogenicity in terms of percentage of subjects with hSBA ≥1:5 and hSBA ≥1:8 at 12 months after two catch up doses previously administered to children at either 12 and 14 or 13 and 15 months of age and 6 months after a booster dose of rMenB+OMV NZ administered at 26 or 27 months of age.
  Both the groups received MMRV at 12 months of age.
Time Frame: 6month post booster dose and 12 months post two catch-up dose vaccination.
Population: Analysis was done on MITT population (Secondary).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B13_15_27 | B12_14_26 | B12+B13Tot
Number analyzed (Participants) | 67 | 18 | 85
Percentage of subjects
  H44/76-SL (hSBA ≥1:5) (12months) | 75 [63 to 84] | 56 [31 to 78] | 71 [60 to 80]
  5/99 (hSBA ≥1:5) (12months) (N= 67, 18, 85) | 97 [90 to 100] | 94 [73 to 100] | 96 [90 to 99]
  NZ98/254 (hSBA ≥1:5) (12months) (N= 67, 18, 85) | 18 [10 to 29] | 6 [0 to 27] | 15 [8 to 25]
  M10713 (hSBA ≥1:5) (12months) (N= 64, 18, 82) | 39 [27 to 52] | 28 [10 to 53] | 37 [26 to 48]
  H44/76-SL (hSBA ≥1:5) (6months) (N= 67, 17, 84) | 99 [92 to 100] | 100 [80 to 100] | 99 [94 to 100]
  5/99 (hSBA ≥1:5) (6months) (N= 67, 18, 84) | 100 [95 to 100] | 100 [80 to 100] | 100 [96 to 100]
  NZ98/254 (hSBA ≥1:5) (6months) (N= 67, 18, 84) | 73 [61 to 83] | 82 [57 to 96] | 75 [64 to 84]
  M10713 (hSBA ≥1:5) (6months) (N= 66, 16, 82) | 92 [83 to 97] | 94 [70 to 100] | 93 [85 to 97]
  H44/76-SL (hSBA ≥1:8) (12months) (N= 67, 18, 85) | 63 [50 to 74] | 56 [31 to 78] | 61 [50 to 72]
  5/99 (hSBA ≥1:8) (12months) (N= 67, 18, 85) | 96 [87 to 99] | 94 [73 to 100] | 95 [88 to 99]
  NZ98/254 (hSBA ≥1:8) (12months) (N= 67, 18, 85) | 15 [7 to 26] | 6 [0 to 27] | 13 [7 to 22]
  M10713 (hSBA ≥1:8) (12months) (N= 64, 18, 82) | 27 [16 to 39] | 22 [6 to 48] | 26 [17 to 36]
  H44/76-SL (hSBA ≥1:8) (6months) (N=67, 17, 84) | 91 [82 to 97] | 100 [80 to 100] | 93 [85 to 97]
  5/99 (hSBA ≥1:8) (6months) (N= 67, 17, 84) | 100 [95 to 100] | 94 [71 to 100] | 99 [94 to 100]
  NZ98/254 (hSBA ≥1:8) (6months) (N= 67, 17, 84) | 52 [40 to 65] | 65 [38 to 86] | 55 [44 to 66]
  M10713 (hSBA ≥1:8) (6months) (N= 66, 16, 82) | 86 [76 to 94] | 81 [54 to 96] | 85 [76 to 92]

6. Secondary Outcome: Percentage of Subjects With at Least Four Fold Increase in hSBA Titers to Evaluate Antibody Response 1 Month Post Booster Dose of rMenB+OMV NZ Vaccination.
Description: To assess the immunogenicity in terms of percentage of subjects with at least four fold increase in hSBA titers 1 month post booster dose of rMenB+OMV NZ administered at 26 or 27 months of age, in children previously administered two catch-up doses of rMenB+OMV NZ at either 12 and 14 or 13 and 15 months of age.Both the groups received MMRV at 12 months of age.
Time Frame: 1 month post booster dose versus prebooster.
Population: Analysis was done on MITT population (Secondary).
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | B13_15_27 | B12_14_26 | B12+B13Tot
Number analyzed (Participants) | 67 | 18 | 85
Percentage of Subjects
  H44/76-SL (N= 66, 18, 84) | 100 [95 to 100] | 100 [81 to 100] | 100 [96 to 100]
  5/99 (N= 67, 18, 85) | 99 [92 to 100] | 100 [81 to 100] | 99 [94 to 100]
  NZ98/254 (N= 65, 18, 83) | 97 [89 to 100] | 94 [73 to 100] | 96 [90 to 99]
  M10713 (N= 62, 16, 78) | 82 [70 to 91] | 88 [62 to 98] | 83 [73 to 91]

7. Secondary Outcome: GMCs to Assess Antibody Persistence at One Year After Two Catch-up Doses and 6 Months After Booster of rMenB+OMV NZ Vaccination Against 287-953 Strain.
Description: To assess the immunogenicity in terms of GMCs determined by ELISA at 12 months after two catch up doses previously administered to children at either 12 and 14 or 13 and 15 months of age and 6 months after a booster dose of rMenB+OMV NZ administered at 26 or 27 months of age.
  Both the groups received MMRV at 12 months of age.
Time Frame: 12 months post two catch-up dose vaccination and 6 months post booster dose.
Population: Analysis was done on MITT population (Secondary).
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration IU/mL
Arm/Group | B13_15_27 | B12_14_26 | B12+B13Tot
Number analyzed (Participants) | 67 | 18 | 85
Concentration IU/mL
  287-953 (6months) (N=67, 17, 84) | 2314 [1596 to 3355] | 3259 [1859 to 5712] | 2597 [2104 to 3205]
  287-953 (12months) | 219 [149 to 322] | 246 [138 to 437] | 227 [185 to 278]

8. Secondary Outcome: GMTs to Characterize Antibody Response at 1 Month and 6 Month Post Two Catch-up Doses of rMenB+OMV NZ Administered to Naive Children at 24 and 26 Months of Age.
Description: To assess the immunogenicity in terms of GMTs through antibody response at 1 month and 6 month post two catch-up doses of rMenB+OMV NZ administered to naive children at 24 and 26 months of age.
Time Frame: 1 month and 6 months post two catch-up doses.
Population: Analysis was done on MITT population (Secondary).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B_24_26
Number analyzed (Participants) | 108
Titers
  H44/76-SL (1months) (N= 105) | 220 [186 to 261]
  5/99 (1months) (N= 103) | 455 [372 to 556]
  NZ98/254 (1months) (N=108 ) | 27 [23 to 32]
  M10713 (1months) (N=100) | 38 [32 to 45]
  H44/76-SL (6months) (N=104) | 22 [18 to 27]
  5/99 (6months) (N= 104) | 71 [57 to 89]
  NZ98/254 (6 months) (N= 104) | 1.88 [1.57 to 2.26]
  M10713 (6months) (N= 104) | 8.04 [6.39 to 10]

9. Secondary Outcome: Percentage of Subjects With hSBA ≥1:5 and hSBA ≥1:8 to Assess Antibody Response at 1 Month and 6 Month Post Two Catch-up Doses of rMenB+OMV NZ Administered to Naive Children at 24 and 26 Months of Age.
Description: To assess the immunogenicity in terms of percentage of subjects with hSBA ≥1:5 and hSBA ≥1:8 through antibody response at at 1 month and 6 month post two catch-up doses of rMenB+OMV NZ administered to naive children at 24 and 26 months of age.
Time Frame: 1 month and 6 months post two catch-up doses.
Population: Analysis was done on MITT population (Secondary)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B_24_26
Number analyzed (Participants) | 108
Percentage of subjects
  H44/76-SL (hSBA ≥1:5) (1months) (N=105) | 100 [97 to 100]
  5/99 (hSBA ≥1:5) (1months) (N= 103) | 99 [95 to 100]
  NZ98/254 (hSBA ≥1:5) (1months) (N= 108) | 98 [93 to 100]
  M10713 (hSBA ≥1:5) (1months) (N= 100) | 97 [91 to 99]
  H44/76-SL (hSBA ≥1:5) (6months) (N=104) | 93 [87 to 97]
  5/99 (hSBA ≥1:5) (6months) (N= 104 ) | 96 [90 to 99]
  NZ98/254 (hSBA ≥1:5) (6months) (N= 104) | 18 [11 to 27]
  M10713 (hSBA ≥1:5) (6months) (N= 104) | 70 [60 to 79]
  H44/76-SL (hSBA ≥1:8) (1months) (N=105) | 100 [97 to 100]
  5/99 (hSBA ≥1:8) (1months) (N= 103) | 99 [95 to 100]
  NZ98/254 (hSBA ≥1:8) (1months) (N= 108) | 96 [91 to 99]
  M10713 (hSBA ≥1:8) (1months) (N= 100) | 95 [89 to 98]
  H44/76-SL (hSBA ≥1:8) (6months) (N=104) | 88 [80 to 93]
  5/99 (hSBA ≥1:8) (6months) (N= 104) | 96 [90 to 99]
  NZ98/254 (hSBA ≥1:8) (6months) (N= 104) | 12 [6 to 19]
  M10713 (hSBA ≥1:8) (6months) (N= 104) | 52 [42 to 62]

10. Secondary Outcome: Percentage of Subjects With Four Fold Increase in hSBA to Assess Antibody Response at 1 Month Post Two Catch-up Doses of rMenB+OMV NZ Administered to Naive Children at 24 and 26 Months of Age.
Description: To assess the immunogenicity in terms of percentage of subjects with fourfold increases in hSBA titers at 1 month post two catch-up doses of rMenB+OMV NZ in children previously administered to naive children at 24 and 26 months of age against 4 strains.
  Analysis was done on MITT population (Secondary).
Time Frame: 1 month post two catch-up doses versus prevaccination
Population: Analysis was done on MITT population (Secondary).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B_24_26
Number analyzed (Participants) | 108
Percentage of subjects
  H44/76-SL (N=105) | 100 [97 to 100]
  5/99 (N= 101) | 99 [95 to 100]
  NZ98/254 (N=108 ) | 96 [91 to 99]
  M10713 (N= 99) | 85 [76 to 91]

11. Secondary Outcome: GMCs to Assess Antibody Response at 1 Month and 6 Month Post Two Catch-up Doses of rMenB+OMV NZ Administered to Naive Children at 24 and 26 Months of Age Against 287-953 Strain.
Description: To assess the immunogenicity in terms of GMCs to assess through antibody response at 1 month and 6 month post two catch-up doses of rMenB+OMV NZ administered to naive children at 24 and 26 months of age against 287-953 strain.
  Analysis was done on MITT population (Secondary).
Time Frame: 1 month and 6 months post two catch-up doses.
Population: Analysis was done on MITT population (Secondary).
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration IU/mL
Arm/Group | B_24_26
Number analyzed (Participants) | 108
Concentration IU/mL
  287-953 strain (1months) | 5448 [4630 to 6411]
  287-953 strain (6months) | 383 [319 to 459]

12. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events (AEs) After Receiving a Booster (Third) Dose of rMenB+OMV NZ Administered at One Year After Two Catch-up Doses of rMenB+OMV NZ, Previously Administered to Children.
Description: To assess the safety and tolerability by reporting solicited local and systemic AEs of a booster (third) dose of rMenB+OMV NZ administered at one year after two catch-up doses of rMenB+OMV NZ, previously administered to children at either 12 and 14 or 13 and 15 months of age in study V72P13E1.
Time Frame: Up to 7 days after any vaccination.
Measure: Number; unit: Number of subjects
Groups:
- B13_15_27: Subjects assessed for safety and tolerability after receiving a booster (third) dose of rMenB+OMV NZ at one year after two catch-up doses of rMenB+OMV NZ, previously administered to children at 13 and 15 months of age.
- B12_14_26: Subjects assessed for safety and tolerability after receiving a booster (third) dose of rMenB+OMV NZ at one year after two catch-up doses of rMenB+OMV NZ, previously administered to children at 12 and 14 months of age.
Arm/Group | B13_15_27 | B12_14_26
Number analyzed (Participants) | 67 | 18
Number of subjects
  Any Local | 64 | 16
  Tenderness (N=67,17) | 63 | 16
  Erythema (N=) | 47 | 13
  Induration | 37 | 9
  Swelling | 35 | 9
  Any Systemic | 53 | 15
  Change Eat. Habits (N=67,17) | 25 | 9
  Sleepiness | 22 | 7
  Vomiting | 4 | 0
  Diarrhea | 4 | 1
  Irritability | 40 | 14
  Unusual Crying | 16 | 5
  Rash | 1 | 0
  Fever ( >= 38C ) | 22 | 6
  Temperature (>= 40 C) | 0 | 0
  Medical Attend. Fever | 0 | 0
  Antipyr. Med. Used Prev | 55 | 12
  Antipyr. Med. Used Trt | 47 | 11

13. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving a Booster (3rd) Dose of rMenB+OMV NZ Administered at One Year After Two Catch-up Doses of rMenB+OMV NZ, Previously Administered to Children.
Description: To assess the safety and tolerability in terms of number of subjects reporting unsolicited adverse events in yerms of serious adverse events (SAEs), atleast possibly related SAEs and AEs leading to withdrawl of a booster (third) dose of rMenB+OMV NZ administered at one year after two catch-up doses of rMenB+OMV NZ, previously administered to children at either 12 and 14 or 13 and 15 months of age in study V72P13E1.
Time Frame: Up to 7 days after any vaccination.
Population: The analysis was done on safety subset.
Measure: Number; unit: Number of Subjects
Arm/Group | B13_15_27 | B12_14_26
Number analyzed (Participants) | 67 | 18
Number of Subjects
  Any AE | 45 | 10
  SAEs | 2 | 1
  At least possibly related SAEs | 0 | 0
  AEs leading to withdrawal | 0 | 0

14. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Two Catch-up Doses of rMenB+OMV NZ Administered to Naive Children at 24 and 26 Months of Age.
Description: To assess the safety and tolerability by reporting solicited local and systemic adverse events of two catch-up doses of rMenB+OMV NZ administered to naive children at 24 and 26 months of age.
Time Frame: Up to 7 days after any vaccination.
Population: The analysis was done on safety subset.
Measure: Number; unit: Number of subjects
Arm/Group | B_24_26
Number analyzed (Participants) | 112
Number of subjects
  Any Local | 110
  Tenderness | 109
  Erythema | 103
  Induration | 75
  Swelling | 58
  Any Systemic | 98
  Change Eat. Habits | 53
  Sleepiness | 70
  Vomiting | 14
  Diarrhea | 23
  Irritability | 84
  Unusual Crying | 47
  Rash | 14
  Fever ( >= 38C) | 44
  Temperature (>= 40 C) | 1
  Medical Attend. Fever | 2
  Antipyr. Med. Used Prev | 33
  Antipyr. Med. Used Trt | 38

15. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving Two Catch-up Doses of rMenB+OMV NZ Administered to Naive Children at 24 and 26 Months of Age.
Description: To assess the safety and tolerability in terms of number of subjects reporting unsolicited adverse events after receiving two catch-up doses of rMenB+OMV NZ administered to naive children at 24 and 26 months of age. The analysis was done on safety subset.
Time Frame: Up to 7 days after any vaccination
Population: The analysis was done on safety subset.
Measure: Number; unit: Number of Subjects
Arm/Group | B_24_26
Number analyzed (Participants) | 112
Number of Subjects
  Any AE | 96
  Serious AEs | 6
  At least possibly related SAEs | 0
  AEs leading to withdrawal | 1

ADVERSE EVENTS:
Time Frame: Throughout the study (solicited and unsolicited from Day 1 to Day 209). Any solicited and unsolicited adverse events, unsolicited SAE, medically attended AEs, AEs leading to withdrawal from the study were collected from day 1 through day.
Description: Any solicited and unsolicited adverse events were reported up to day 7 post vaccination for group B13_15_27, B12_14_26 and B_24_26 . Since no vaccination was administered to group B246_12M12 and B246_12M13 and antibody persistence was explored at 12 months after the fourth dose rMenB+OMV NZ, the two group are excluded from the reporting AEs.
Groups:
- B12_14_26: Subjects assessed for safety and tolerability after receiving a booster (third) dose of rMenB+OMV NZ at one year after two catch-up doses of rMenB+OMV NZ, previously administered to children at either 12 and 14 months of age.
- B24_26: Subjects assessed for safety and tolerability after two catch-up doses of rMenB+OMV NZ administered to naive children at 24 and 26 months of age.
Arm/Group | B13_15_27 | B12_14_26 | B24_26
Serious Adverse Events (participants affected / at risk) | 2/67 | 1/18 | 6/112
Other Adverse Events (participants affected / at risk) | 67/67 | 18/18 | 110/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B13_15_27 (N=67) | B12_14_26 (N=18) | B24_26 (N=112)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenoidal Hypertrophy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 1
Pneumonia Respiratory Syncytial (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B13_15_27 (N=67) | B12_14_26 (N=18) | B24_26 (N=112)
Somnolence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 7 | 70
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 14
Speech Disorder Developmental (Nervous system disorders) | 0 | 1 | 0
Crying (General disorders) | 16 | 5 | 47
Induration (General disorders) | 1 | 1 | 4
Injection Site Erythema (General disorders) | 47 | 13 | 103
Injection Site Pain (General disorders) | 63 | 16 | 109
Injection Site Swelling (General disorders) | 35 | 9 | 58
Pyrexia (General disorders) | 22 | 6 | 46
Tenderness (General disorders) | 1 | 1 | 0
Eating Disorder (Psychiatric disorders) | 25 | 9 | 53
Irritability (Psychiatric disorders) | 40 | 14 | 84
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 24
Vomiting (Gastrointestinal disorders) | 4 | 0 | 15
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 18
Bronchitis (Infections and infestations) | 4 | 1 | 14
Conjunctivitis (Infections and infestations) | 5 | 0 | 16
Ear Infection (Infections and infestations) | 1 | 0 | 6
Exanthema Subitum (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 6
Nasopharyngitis (Infections and infestations) | 5 | 2 | 9
Otitis Media (Infections and infestations) | 7 | 1 | 18
Pharyngitis (Infections and infestations) | 2 | 0 | 9
Pneumonia (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 8
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 1 | 20
Viral Infection (Infections and infestations) | 7 | 1 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.